CLINICAL TRIAL: NCT06263660
Title: Exploratory Randomized, Placebo-Controlled, Double-Blind Study to Evaluate the Effect of a Keto-Like Supplement in Depressed Patients on Functional Brain Responses to Positive and Negative Stimuli
Brief Title: Evaluation of a Keto-Like Supplement on Brain Responses to Emotional Stimuli in Depression
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Laureate Institute for Brain Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2022-007
Record Dates: First submitted 2024-02-05; First posted 2024-02-16 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Keto-like supplement (Active Comparator): Participants will receive standardized 9.25g stick packs of the keto-like supplement. The study participants will take one of these stick packs dissolved in water three times a day (morning, noon, and evening) for 8 weeks.
  Interventions: Dietary Supplement: Keto-like supplement
- Placebo (Placebo Comparator): Participants will receive standardized 9.25g stick packs of placebo. The study participants will take one of these stick packs dissolved in water three times a day (morning, noon, and evening) for 8 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Keto-like supplement — Participants will consume 9.25g stick packs of the keto-like supplement dissolved in water 3 times per day for 8 weeks.
  Arms: Keto-like supplement
Dietary Supplement: Placebo — Participants will consume 9.25g stick packs of placebo dissolved in water 3 times per day for 8 weeks.
  Arms: Placebo

SUMMARY:
This study aims to determine whether a keto-like supplement relative to placebo results in functional brain changes during fMRI tasks evaluating positive and negative valence in individuals with moderate to severe depression. In this double-blind randomized placebo-controlled trial, 75 individuals with a Patient Health Questionnaire (PHQ-9) scale score ≥ 10 (MDD) will be enrolled to participate in an 8-week treatment study to obtain 60 completers. Participants will be randomized with a 1-1 ratio to receive the keto-like supplement (n= 30 completers) or placebo (n=30 completers) taken orally three times per day for 8 weeks. Participants will undergo a 10.5-hour screening/baseline evaluation visit split over 2 days at week 0 including questionnaires, neuroimaging before and after supplement or placebo administration and blood draws, office visits at week 2 (1.5 hours), week 4 (3 hours), week 6 (0.5 hours), week 8 (6 hours), a follow-up visit at week 10 (1.5 hours) and two phone calls between visits (weeks 1 and 3) during which a brief clinical assessment will be obtained (10 minutes each). The total time involved in the study is approximately 23.5 hours.

ELIGIBILITY:
Inclusion Criteria:

* Meets the Diagnostic and statistical manual - 5 (DSM-5) diagnostic criteria for MDD without psychotic features (past or present), as confirmed by the M.I.N.I v7.0
* PHQ-9 score of ≥10
* C-Reactive Protein (CRP) value > 1
* Age 18-65
* Consent ability and written consent
* Body Mass Index (BMI) between 19 and 38 kg/m2
* Medically stable based on clinical laboratory tests, medical history and vital signs
* No intention to become pregnant during the study
* A woman of childbearing potential must have a negative serum pregnancy test at screening
* Consent that possible random finding is reported (e.g. brain abnormality during imaging)

Exclusion Criteria:

* Has a current or recent history of clinically significant suicidality
* Has a history of moderate or severe substance or alcohol use disorder according to DSM-5 criteria, except nicotine or caffeine, within 12 months before screening
* Has positive test result(s) for alcohol or drugs of abuse (including methadone, opiates, cocaine, cannabinoids, amphetamine/methamphetamine and ecstasy)
* Has a current diagnosis of a psychotic disorder (e.g. schizophrenia, bipolar disorder), an eating disorder (e.g. anorexia, bulimia), or learning disability or a personality disorder that is considered by the investigator to interfere with the ability of the subject to adhere to the protocol (e.g. narcissistic personality, borderline personality disorder)
* Change in medication dose and/or frequency within the last 6 weeks. Participants must be on stable medications for 6 weeks prior to enrollment.
* Plans to change medication dose/frequency during the course of the study. Must plan to remain on stable dose for the duration of the study, unless otherwise indicated by their provider during the course of the study.
* Plans to take vitamins and/or mineral supplements during the study. Must refrain for the duration of the study
* Unable to complete MRI scans
* Is a woman who is pregnant or breast feeding
* Plans to conceive a child while enrolled in this study or within 3 months after the last dose of the keto-like supplement
* Has received an investigational drug/vaccines, used an invasive investigational medical device within 60 days before the planned first dose of the keto-like supplement or has participated in 2 or more interventional clinical studies in the previous 1 year, or is currently enrolled in any drug or non-drug interventional study.
* Has had major surgery, (i.e. requiring general anesthesia) within 12 weeks before screening, or will not have fully recovered from surgery, or has surgery planned during the time they are expected to participate in the study.
* Intake of Omega 3 fatty acids (DHA, EPA, fish oil supplements)
* Significant cognitive impairment, clinically relevant or progressive disease (e.g., liver, kidney, cardiovascular system, respiratory tract, vascular system, brain, metabolism, thyroid) that could affect the course of the study
* Known metabolic disorders (e.g., fatty acid oxidation disorders, ketolysis/ketogenesis or glucogenesis disorder, hyperinsulinism (e.g., pancreatic neuroendocrine tumor), pyruvate carboxylase deficiency, Type 1 and Type 2 diabetes
* Allergy to Stevia sweetener, malic acid or orange flavoring
* Concern for inability to maintain adherence to the keto-like supplement administration protocol
* Currently practicing a ketogenic or paleo diet or planning to do so during the study period.
* Change in body weight of more than 5 kg within one month before the start of the intervention
* Medical, psychiatric or other conditions that restrict the patient's following abilities: to interpret the study information, to give informed consent, to adhere to the rules of the protocol, or to complete the study
* Contraindications to MRI examinations [persons with metallic implants (e.g., intracranial metal clips) and carriers of electronic devices (e.g., pacemaker) or persons with claustrophobia]

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-01-09 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
BOLD response during Monetary Incentive Delay Task | week 0 pre, week 0 post, week 8
  P5vP0 contrast in the nucleus accumbens during the Monetary Incentive Delay Task

SECONDARY OUTCOMES:
BOLD response during Adjective Task | week 0 pre, week 0 post, week 8
  SELFvWORD contrast in the medial prefrontal cortex during the Adjective task

CONTACTS AND LOCATIONS:
Overall Officials: Martin Paulus, MD, Principal Investigator — Laureate Institute for Brain Research
Locations (1):
- Laureate Institute for Brain Research, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No